CLINICAL TRIAL: NCT06195631
Title: Evaluating the SCOPE-E Bundle, a Standardized Checklist Bundle for Optimizing Procedural Ergonomics in Endoscopy: An Effectiveness-Implementation Cluster Randomized Trial
Brief Title: Evaluating a Standardized Checklist Bundle for Optimizing Procedural Ergonomics in Endoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Study had not been IRB approved, no one took over the study, and PI moved to another institution.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PAWA SCOPE-E Bundle
Record Dates: First submitted 2023-12-22; First posted 2024-01-08 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2025-08

CONDITIONS: Injuries
Keywords: Ergonomics; Endoscopy related injury ( ERI); Checklist
MeSH Terms: conditions — Wounds and Injuries | interventions — Endoscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE- E) Bundle (Experimental): Endoscopists in each unit that is randomized to the intervention will be asked to use an ergonomic check list to conduct a verbal time-out before commencing each colonoscopy procedure.
  Interventions: Behavioral: Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE- E) Bundle
- Standard of practice (No Intervention): Usual practice does not involve any of the core components of the SCOPE-E bundle. Endoscopy units in the control arm will not undergo any targeted intervention(s) to enhance ergonomic behaviors throughout the study period.

INTERVENTIONS:
Behavioral: Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE- E) Bundle — The SCOPE-E bundle is a multicomponent intervention designed to improve endoscopy ergonomics. The bundle is composed of one core intervention and 5 evidence-based implementation strategies which are defined as methods to enhance the adoption, implementation and sustainment of the core intervention. The core intervention is a pre-endoscopy ergonomic time-out checklist. The implementation strategies are endoscopist education, checklist documentation, visual reminders, nursing engagement and leadership support.
  Arms: Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE- E) Bundle

SUMMARY:
The goal of this Hybrid Type 2 effectiveness-implementation trial is to test the Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE-E) bundle-a multicomponent intervention comprised of a pre-procedure ergonomic timeout checklist and evidence-based implementation strategies-as a strategy to mitigate the risk of Endoscopy-related injuries (ERI) during colonoscopy.

DETAILED DESCRIPTION:
Endoscopy-related injuries (ERI) occur frequently, emphasizing the crucial need to integrate ergonomic principles into endoscopic practice to mitigate risks and prioritize the health and well-being of endoscopists. Checklists are a proven strategy in healthcare behavior modification; however, the efficacy of a pre-procedure ergonomic timeout checklist remains underexplored. To bridge this gap, the aim is to evaluate the effectiveness and implementation of the Standardized Checklist for Optimizing Procedural Ergonomics in Endoscopy (SCOPE-E) bundle-a multicomponent intervention comprised of a pre-procedure ergonomic timeout checklist and evidence-based implementation strategies-as a strategy to mitigate the risk of ERI during colonoscopy.

Conducted will be a Hybrid Type 2 cluster randomized controlled trial across 10 endoscopy units in North America with 100 participants. Units will be randomized to the SCOPE-E bundle or usual practice. Effectiveness will be measured by comparing Rapid Entire Body Assessment (REBA) scores before and 3 months after implementation between intervention and control groups. Simultaneously, implementation outcomes will be assessed to understand the practicality of this ergonomic intervention and inform widescale adoption. If demonstrated to be effective, the SCOPE-E Bundle is a feasible and cost-effective intervention that holds significant promise for improving ergonomics globally.

ELIGIBILITY:
Inclusion Criteria:

* Endoscopists who perform colonoscopy at least once per week at one of the participating endoscopy units and who are willing to sign an informed consent form before any study procedures are performed

Exclusion Criteria:

* Endoscopists-in-training will be excluded as will endoscopy units that do not have adjustable monitors and patient beds

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01 (Estimated); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Difference in mean Rapid Entire Body Assessment (REBA) scores during colonoscopy between groups (intervention and control) - assessed using ErgoGENIUS (an artificial intelligence posture analysis program) | Month 3
  REBA, a validated measure of entire body ergonomics which considers joint positioning, force exertion, repetitive movements and postural shifts, is a surrogate for Endoscopic Related Injury (ERI) risk. The minimum REBA Score = 1, and the maximum REBA Score = 15. The design goal for the REBA assessment is a score of 4

SECONDARY OUTCOMES:
Difference in the percentage of time endoscopists spend during colonoscopy in postures at medium, high or very high risk of ERI (i.e., REBA score >4). | Month 3
  REBA, a validated measure of entire body ergonomics which considers joint positioning, force exertion, repetitive movements and postural shifts, is a surrogate for Endoscopic Related Injury (ERI) risk. The minimum REBA Score = 1, and the maximum REBA Score = 15. The design goal for the REBA assessment is a score of 4
Reach - Number of endoscopists per unit who consent to participate | Month 3
  Number of endoscopists per unit who consent to participate.
Adoption - Percentage of colonoscopies | Baseline and Month 3
  Percentage of colonoscopies where a pre-endoscopy ergonomic timeout is completed over a 1-week period pre- and 3-months post intervention initiation.
Feasibility - time taken to complete the endoscopy ergonomic timeout | Month 3
  Mean time taken to complete the endoscopy ergonomic timeout, measured over 1-week period 3-months post-intervention initiation.
Fidelity - Rate of inclusion of all checklist components in the pre-endoscopy timeout | Month 3
  Rate of inclusion of all checklist components in the pre-endoscopy timeout, number and source of interruptions during timeout, and rate of checklist documentation, measured over 1-week period 3-months post-intervention initiation.
Acceptability - Survey Score | Month 3
  Endoscopists' and nurses ± technicians' perceived acceptability of the SCOPE-E bundle (numerical rating, data source: post-implementation survey. Scores range from 0-7 with higher scores meaning more acceptance
Adaptation - Survey Score | Month 3
  Self-reported adaptations by endoscopists to make the SCOPE-E bundle fit to their context (qualitative data, data source: post-implementation survey).Scores range from 0-7 with higher scores meaning more adaptation
Sustainability - Survey Score | Month 3
  Intention to continue implementation beyond study period (numerical rating, source: post- survey). Scores range from 0-7 with higher scores meaning more sustainability

CONTACTS AND LOCATIONS:
Overall Officials: Pawa Swati, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No